CLINICAL TRIAL: NCT01910766
Title: Combined Coenzyme Q10 and Clomiphene Citrate (CC) for Ovulation Induction in CC-resistant Patients With Polycystic Ovary Syndrome
Brief Title: Coenzyme Q10 and Clomiphene Citrate (CC) for Ovulation Induction in Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, ahmed M. badawy, Professor of Obstetrics & Gynecology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CoQ10
Record Dates: First submitted 2013-07-19; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: pcos; coenzymeQ10; clomiphene citrate
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — coenzyme Q10; Clomiphene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coenzyme Q10/CC group (Experimental): Intervention:
  Coenzyme Q10 (CoQ10) and clomiphene citrate group (55 patients, 82 cycles) Patients in CoQ10/CC group took CC (Global Napi, Cairo, Egypt) 100 mg/day from cycle days 2-6, and CoQ10 Mepaco, Enshas Elraml, Sharkhia, Egypt), in a dose of 60 mg 3 times day capsules orally starting on cycle day 2 and continued till the day of human chorionic gonadotropin (hCG) administration
  Interventions: Drug: Coenzyme Q10; Drug: clomiphene citrate
- CC alone group (Active Comparator): Intervention:
  CC (Global Napi, Cairo, Egypt) 100 mg/day from cycle days 2-6
  Interventions: Drug: clomiphene citrate

INTERVENTIONS:
Drug: Coenzyme Q10 — no more details
  Other Names: CC 100 mg/day 2-6 and CoQ10,60 mg 3 times day orally on day 2 till hCG
  Arms: Coenzyme Q10/CC group
Drug: clomiphene citrate

SUMMARY:
Objective of the study was to evaluate the effect of combination of oral Coenzyme Q10 (CoQ10), with clomiphene citrate (CC) for ovulation induction in CC-resistant polycystic ovary syndrome (PCOS).In a prospective controlled randomized trial performed in a university hospital and private practice setting. One hundred ten infertile women with PCOS resistant to CC were randomized to either combined CC/CoQ10 (51 patients, 82 cycles) or CC 150 mg/day alone (50 patients, 71 cycles) for ovulation induction in patients with CC-resistant PCOS.

Main outcome measures: Number of follicles, serum E2, serum P, endometrial thickness, pregnancy rate (PR) and miscarriage rate.

DETAILED DESCRIPTION:
No more details

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS based on the revised 2003 consensus on diagnostic criteria and long-term health risks related to PCOS (2003).
* All women were previously treated with 100 mg of CC daily for 5 days per cycle, for two to three cycles with persistent anovulation or ovulate with very thin endometrium <5 mm at the time of hCG administration

Exclusion Criteria:

* patients with hyperprolactinaemia,
* hypercorticism and
* thyroid dysfunction.
* patients receiving medications as cholesterol lowering drugs, as statins, beta-blockers, and tricyclic antidepressants

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of ovulating patients | 1-2 months

SECONDARY OUTCOMES:
Number of pregnancies | 1-2 months

OTHER OUTCOMES:
Number of miscarriages | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Derived] El Refaeey A, Selem A, Badawy A. Combined coenzyme Q10 and clomiphene citrate for ovulation induction in clomiphene-citrate-resistant polycystic ovary syndrome. Reprod Biomed Online. 2014 Jul;29(1):119-24. doi: 10.1016/j.rbmo.2014.03.011. Epub 2014 Mar 26. PMID 24813752